CLINICAL TRIAL: NCT05166187
Title: Best Practice Advisory to Initiate High-Intensity Statin Therapy in Patients With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Aaron W. Aday, MD, MSc, Assistant Professor, Division of Cardiovascular Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 212294
Record Dates: First submitted 2021-12-06; First posted 2021-12-21 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Statin; Electronic alert; Best Practice Advisory
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to the intervention arm will have a Best Practice Advisory (BPA) displayed as part of the discharge order workflow. This BPA requires clinicians to choose an option before completing the discharge documentation. Options include ordering one of the appropriate statins or documenting that the medication is contraindicated, the patient declined, or the patient does not meet criteria for a high-intensity statin.
  Interventions: Other: Best Practice Advisory
- Usual Care (No Intervention): Patients randomized to the usual care arm will have the identical set of windows displayed in the discharge workflow minus the BPA window.

INTERVENTIONS:
Other: Best Practice Advisory — Patients in this arm will have a Best Practice Advisory displayed in the Electronic Medical Record (EMR) as part of the discharge order workflow.
  Arms: Intervention

SUMMARY:
The purpose of this study is to understand how a Best Practice Advisory (BPA) for high-intensity statin therapy in patients with Peripheral Artery Disease impacts prescription rates.

DETAILED DESCRIPTION:
The central hypothesis is that an automated best practice advisory embedded within the electronic medical record (EMR) will improve prescription of high-intensity statins among hospitalized patients with Peripheral Artery Disease (PAD).

Aim 1: To assess the impact of an automated best practice advisory, deployed as part of the standard hospital discharge workflow within the electronic medical record, on high-intensity statin prescription among hospitalized patients with PAD.

Aim 2: To assess the impact of an automated best practice advisory, deployed as part of the standard hospital discharge workflow within the electronic medical record, on short-term cardiovascular outcomes among hospitalized patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

* Primary hospital diagnosis of PAD defined by ICD/CPT codes
* Inpatient status at the adult hospital at Vanderbilt University Medical Center
* Not currently prescribed a high-intensity statin (atorvastatin 40-80mg daily or rosuvastatin 20-40mg daily)

Exclusion Criteria:

* On comfort measures
* History of statin allergy or intolerance recorded in the EMR
* History of rhabdomyolysis defined by International Classification of Diseases/Current Procedural Terminology (ICD/CPT) codes
* History of hepatitis A, B, or C defined by ICD/CPT codes
* Pregnant
* Aspartate aminotransferase >120 units/L within 30 days of alert
* Alanine aminotransferase >165 units/L within 30 days of alert
* Primary hospital diagnosis of acute myocardial infarction defined by ICD/CPT codes
* Primary hospital diagnosis of acute stroke defined by ICD/CPT codes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-08-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Frequency of High-Intensity Statin Prescription at discharge | Baseline, upon patient discharge through study completion, average of six months
  Frequency will be measured by identifying the number of high-intensity statin prescriptions at discharge
Frequency of High-Intensity Statin Prescription at 90 days post-discharge | 90 days post-discharge
  Frequency will be measured by identifying the number of high-intensity statin prescriptions at 90 days post-discharge.

SECONDARY OUTCOMES:
Frequency of a Composite of Cardiovascular Events | Baseline, upon patient discharge to 90 days post-discharge through study completion
  Frequency will be measured by identifying the number of cardiovascular events including myocardial infarction, coronary revascularization, stroke, lower extremity arterial revascularization, or all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron W Aday, MD, MSc, Principal Investigator — VUMC Cardiovascular Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States